CLINICAL TRIAL: NCT04347694
Title: COVID-19 Serology in Nephrology Health Care Workers
Brief Title: Study to Determine the Immunization Status Among Nephrological Health Care Personnel Against SARS-CoV-2 in a Single Center Over the Course of 12 Months During the Worldwide COVID-19 Pandemic.
Acronym: CONEC
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Dr. Thomas Reiter, Specialist in Internal Medicine, Medical University of Vienna
Other Study IDs: 1357/2020
Record Dates: First submitted 2020-04-12; First posted 2020-04-15 (Actual); Last update posted 2020-09-02 (Actual); Status verified 2020-09

CONDITIONS: SARS-CoV 2; Immunization; Infection
Keywords: Nephrology; SARS-CoV-2; Vienna; Health Care Personnel
MeSH Terms: conditions — Infections

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — blood, urine
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Infections with Corona-Viruses have shown to be a menace for patients with comorbidities such as hypertension, diabetes, cardiovascular disease or immunosuppression. Those are features almost every nephrological patient brings along, especially those on maintenance dialysis and those with renal transplant. Since the emergence of the novel coronavirus SARS-CoV-2 in November 2019 in Mainland China the fear for pandemic infections has increased. But not only is the course of infection itself important, the prevention of transmission to and by attending medical personnel should be put into perspective. Thus there is a lack of sufficient data of occult immunization or persistent state on immunization.

In our study up to 400 health care personnel will be screened serologically for IgM, IgA and IgG against the SARS-CoV-2 virus. Blood and urine samples throughout 12 months will be sampled and analyzed.

The aim of the study is to identify the rate of occult immunization and at the same time to gather data about the persistence of immune response to an infection with SARS-CoV-02. The results will help provide sufficient safety measures for health care providers and renal patients undergoing unavoidable clinical treatment.

ELIGIBILITY:
Inclusion Criteria:

* Health Care Personnel and other staff at the Division of Nephrology & Dialysis at the Medical

Exclusion Criteria:

* Not matching the inclusion criteria

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Health Care Personnel
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2020-04-11 (Actual); Primary Completion 2021-04-11 (Estimated); Study Completion 2021-04-11 (Estimated)

PRIMARY OUTCOMES:
Status of Immunization | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Thomas J Reiter, MD, Principal Investigator — Medical University of Vienna
Locations (1):
- Medical University of Vienna, Division for Nephrology and Dialysis, Vienna, Austria

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Gerges D, Kapps S, Hernandez-Carralero E, Freire R, Aiad M, Schmidt S, Winnicki W, Reiter T, Pajenda S, Schmidt A, Sunder-Plassmann G, Wagner L. Vaccination with BNT162b2 and ChAdOx1 nCoV-19 Induces Cross-Reactive Anti-RBD IgG against SARS-CoV-2 Variants including Omicron. Viruses. 2022 May 28;14(6):1181. doi: 10.3390/v14061181. PMID 35746653
- [Derived] Reiter T, Pajenda S, Wagner L, Gaggl M, Atamaniuk J, Holzer B, Zimpernik I, Gerges D, Mayer K, Aigner C, Strassl R, Jansen-Skoupy S, Fodinger M, Sunder-Plassmann G, Schmidt A. COVID-19 serology in nephrology healthcare workers. Wien Klin Wochenschr. 2021 Sep;133(17-18):923-930. doi: 10.1007/s00508-021-01848-5. Epub 2021 Apr 9. PMID 33835265